CLINICAL TRIAL: NCT06284876
Title: A Multicenter, Double-blind, Randomized, Parallel, Active-controlled, Phase III Clinical Trial to Evaluate the Efficacy and Safety of Ilaprazole 10 mg in Prevention NSAIDs Associated Peptic Ulcer
Brief Title: Study to Evaluate the Efficacy and Safety of Ilaprazole 10 mg in Prevention NSAIDs Associated Peptic Ulcer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Il-Yang Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IY-NTNS03
Record Dates: First submitted 2024-02-21; First posted 2024-02-29 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Peptic Ulcer
MeSH Terms: conditions — Peptic Ulcer | interventions — ilaprazole; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ilaprazole 10 mg (Experimental): Take Ilaprazole 10 mg 1 tablet + Placebo of Lansoprazole 15 mg 1 capsule by mouth, with water, once daily.
  Interventions: Drug: Ilaprazole; Drug: Lansoprazole Placebo
- Lansoprazole 15 mg (Active Comparator): Take Lansoprazole 15 mg 1 capsule + Placebo of Ilaprazole 10 mg 1 tablet by mouth, with water, once daily.
  Interventions: Drug: Lansoprazole; Drug: Ilaprazole Placebo

INTERVENTIONS:
Drug: Ilaprazole — Ilaprazole 10 mg
  Other Names: Noltec(the brand name)
  Arms: Ilaprazole 10 mg
Drug: Lansoprazole — Lansoprazole 15 mg
  Other Names: Lanston(the brand name)
  Arms: Lansoprazole 15 mg
Drug: Ilaprazole Placebo — Placebo of Ilaprazole 10 mg
  Other Names: Ilaprazole Placebo-matching tablet
  Arms: Lansoprazole 15 mg
Drug: Lansoprazole Placebo — Placebo of Lansoprazole 15 mg
  Other Names: Lansoprazole Placebo-matching tablet
  Arms: Ilaprazole 10 mg

SUMMARY:
To demonstrate the non-inferiority of Ilaprazole 10 mg to the active control in prevention of NSAIDs-associated peptic ulcer, as assessed by the proportion of subjects with peptic ulcer by Week 24

DETAILED DESCRIPTION:
Not provided

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and females aged 19 years or older on the day of informed consent
2. Subjects requiring continuous treatment or receiving treatment with NSAIDs
3. Subjects with at least one of following peptic ulcer risk factors at the time of Screening
4. Subjects who have provided voluntary informed consent for the study participation after the study is explained

Exclusion Criteria:

1. Subjects with Gastroesophageal varices, Esophageal stricture or ulcerous stenosis, Gastrointestinal bleeding or perforation, Esophageal dysplasia and else based on the screening EGD results.
2. Subjects with inflammatory bowel diseases, pancreatitis, pyloric obstruction, and primary esophageal motility disorder
3. Subjects with confirmed history of malignancy within 5 years prior to Screening
4. Positive human immunodeficiency virus (HIV) antigen/antibody at Screening

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Ilaprazole, Lansoprazole peptic ulcer | at 24 weeks
  Proportion of subjects with newly developed peptic ulcer until Week 24 after the IP treatment

SECONDARY OUTCOMES:
Ilaprazole, Lansoprazole peptic ulcer | at 12 weeks
  Proportion of subjects with newly developed peptic ulcer until Week 12 after the IP treatment
Ilaprazole, Lansoprazole GI bleeding | at 12, 24 weeks
  Proportion of subjects with upper GI bleeding by Week 12 and Week 24 after the IP treatment

CONTACTS AND LOCATIONS:
Overall Officials: JungSoo Song, M.D., Principal Investigator — Chung-Ang University Hospital Center
Locations (2):
- South Korea (2):
  - Chung Ang University Hospital, Seoul
  - Chung-Ang University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No